CLINICAL TRIAL: NCT01440075
Title: Prevalence and Early Markers of Atherosclerosis in Adults With a History of Kawasaki Disease
Acronym: Kawasaki
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009.593
Record Dates: First submitted 2011-09-21; First posted 2011-09-26 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients KD (Other): Adults with a history of KD disease in childhood
  Interventions: Other: Cardiac evaluation
- Case Control (Other): Control group, healthy volunteers matched for age and sex with the KD group
  Interventions: Other: Cardiac evaluation

INTERVENTIONS:
Other: Cardiac evaluation — complete cardiac evaluation with :
  Electrocardiogram Echodoppler Echodoppler with dobutamine stress Carotid Echodoppler Coronary scan Positron emission tomography with adenosine stress Blood test (search for early atherosclerosis marker Genotyping

SUMMARY:
Kawasaki disease (KD) is an acute systemic vasculitic syndrome with coronary tropism.

It has been reported worldwide, but it is ten times more common in Asian population. The annual incidence in children under 5 years in Europe is estimated at 8 to 100000. It is the second vasculitis of the child by its frequency after rheumatoid purpura. It occurs in 80% of cases between 1 and 5 years, with a maximal incidence around the age of 12 months.

It may results in acquired heart disease in children in developed countries, and may be the cause of premature coronary artery disease in adulthood.

A polymorphism was recently associated with the occurrence of disease in a Japanese and U.S population. (C allele of SNP itpkc_3, with a risk multiplied by 2). However, data are conflicting on this issue and the prevalence of this allel is unknown in North America and Europe populations.

The clinical picture of KD associate a persistent fever and an antipyretics resistance with mucocutaneous signs and bulky cervical lymphadenopathy usually unilateral. Diagnosis is confirmed by the presence of five clinical signs (major criteria). The presence of inconsistent coronary lesions in cardiac ultrasound can confirm the diagnosis.

KD can resolve spontaneously with no treatment. The severity of the disease is primarily related to complications of coronary aneurysms in acute or chronic stages.

Several arguments support the fact that adult patients have diffuse vascular lesions different from aneurysmal lesions initially described in childhood.

Despite abundance of publications on KD, there is no prospective or retrospective study which explored anomalies resulting from KD in adult subjects.

Therefore, this project will describe the patient's vascular evolution, the prevalence of atherosclerotic lesions and to determine the biological and functional abnormalities, markers of accelerated atherosclerosis.

Hypothesis : A history of Kawasaki disease represents a cardiovascular risk factor in adulthood.

The main objective is to evaluate the prevalence of atherosclerotic lesions, their extent and their severity in adults with a history of KD in childhood compared to a control population.

ELIGIBILITY:
Inclusion Criteria:

* History of KD before the age of 18, with or without macroscopic coronary lesions in the childhood phase. (KD group only)
* 18 years old or older at the time of the study.
* Agree on participating to all explorations of the study.
* Accept genotyping.
* Absence of cardiovascular risk factors

Exclusion Criteria:

* Atypical KD (KD group only)
* Documented or suspected coronary ischemia,
* Refusal to participate to the study or sign the consent
* Contra-indication to the injection of iodinated contrast agents (allergy, renal failure)
* Hypersensitivity to dobutamine,
* No effective contraception method for females with child bearing potential,
* Breastfeeding, or pregnant females,
* Treatment modifying endothelial reactivity
* History of severe intolerance to iodinated contrast agents,
* Subjects who can't hold their breath for at least 20 seconds,
* Irregular or absence of sinus rhythm, especially atrial or ventricular arrhythmia
* Unability to give information to the subject,
* No coverage from a Social Security system
* Deprivation of civil rights

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-10-10 (Actual); Primary Completion 2015-04-13 (Actual); Study Completion 2015-04-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of carotid and coronary atherosclerotic plaques at vascular Doppler ultrasound and coronary scan in the KD population versus control population | 1 day

SECONDARY OUTCOMES:
Early markers of atherosclerosis | 1 day
  Secondary Outcomes consist of early markers of atherosclerosis:
  * Carotid intima-media thickness
  * Endothelial dysfunction of coronary arteries,
  * Myocardial blood flow at rest and under pharmacological stress (adenosine)
  * Myocardial systolic function overall and segmental at rest and under pharmacological stress (dobutamine)
  * Early biological markers of atherosclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Di Filippo, Pr, Principal Investigator — Hospices Civiles de Lyon
Locations (1):
- Hopital cardiologique Louis Pradel, Bron, France